CLINICAL TRIAL: NCT07294053
Title: Sugary Drink Labeling Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0901a; R01DK135743 (NIH)
Record Dates: First submitted 2025-12-11; First posted 2025-12-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Added sugar warning (Experimental)
  Interventions: Behavioral: Added sugar warning
- Control label (Other)
  Interventions: Behavioral: Control label

INTERVENTIONS:
Behavioral: Added sugar warning — The added sugar warning will say "High in added sugar." The warning will be in an octagon-shaped label. These warnings will be placed on the front of sugary drink containers in the experimental store.
  Arms: Added sugar warning
Behavioral: Control label — The control label will display a barcode in a square shape. These labels will be placed on the front of sugary drink containers in the experimental store.
  Arms: Control label

SUMMARY:
This study aims to examine the effects of added sugar warning labels on sugary drinks. Participants will be assigned to view either added sugar warning labels or control labels, applied on sugary drinks in an experimental store. Participants will shop for beverages in the store and take a computer survey at 4 visits spaced approximately 1 week apart.

DETAILED DESCRIPTION:
This study aims to determine whether new added sugar warnings on sugary drinks lead to decreased amount of added sugar purchased from sugary drinks. The investigators aim to enroll approximately 543 adults ages 18 and older who have consumed at least one sugary drink in the past week. Participants will attend 4 in-person study visits at the study experimental store, spaced approximately 1 week apart. Participants will be randomized to 1 of 2 trial arms at the time of scheduling. At the first visit, participants will provide written informed consent. At each study visit, participants will shop for beverages in the store and take a computer survey. Participants will view sugary drinks in the store labeled per their trial arm. Researchers will record in-store purchases, and other self-reported measures will be assessed via the computer surveys.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Bought sugary drinks from a store at least once during the past week
* Willing to attend 4 in-person study appointments

Exclusion Criteria:

* Living in the same household as someone else in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 543 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Amount of added sugars purchased from sugary drinks | Assessed once a week for up to 4 weeks, starting on the day of enrollment.
  Measured using purchase data for sugary drinks, defined as drinks that contain at least 20% of the daily value for added sugar. The total amount of added sugars (in grams) in all sugary drinks purchased will be calculated.

SECONDARY OUTCOMES:
Amount of total sugars purchased from all beverages | Assessed once a week for up to 4 weeks, starting on the day of enrollment.
  Measured using purchase data for all drinks. The total amount of total sugars (in grams) in all drinks purchased will be calculated.
Volume of sugary drinks consumed in the past 7 days | Assessed 1 time, approximately 3 weeks after enrollment.
  Measured using survey items adapted from the BEV-Q 15 measure. The survey items assess frequency of consumption of sugary drinks and typical volume of sugary drinks consumed in the past 7 days. Researchers will multiply frequency by typical volume to estimate the total volume of sugary drinks consumed in the past 7 days, reported in fluid ounces.
Intentions to reduce sugary drink consumption | Assessed once a week for up to 4 weeks, starting on the day of enrollment.
  Measured using 3 survey items: 1) "How interested are you in drinking fewer sugary drinks in the next week?" 2) "How much do you plan to drink fewer sugary drinks in the next week?" and 3) "How likely are you to drink fewer sugary drinks in the next week?". Response options are on a 5-point scale with lowest endorsement coded as 1 and highest endorsement coded as 5. Researchers will average responses to the 3 items to create a scale score. Higher scores indicate greater intentions to reduce sugary drink consumption.
Forgoing sugary drinks | Assessed approximately 1 week, 2 weeks, and 3 weeks after enrollment.
  Measured using 5 survey items asking participants how often they chose to forgo sugary drinks during the study (e.g., "In the last 7 days, how often have you stopped yourself from having sugary drinks because you wanted to cut back?"). Response options are on a 5-point scale ranging from "Never" coded as 0, to "10 or more times", coded as 10. Researchers will average responses to the 5 items. Higher scores indicate greater frequency of forgoing sugary drinks.
Learning something new | Assessed once, approximately 3 weeks after enrollment.
  Measured using 1 survey item: "Did you learn something new from the labels?" where response options are "Yes" (coded as 1) and "No" (coded as 0).
Correct identification of beverages high in added sugar | Assessed once, on the day of enrollment.
  The survey will show 6 drinks in random order, asking participants "Is this product high in sugar?" with response options of "No", "Yes", and "Don't know." 4 of the drinks will be high in added sugar and 2 will not be high in added sugar. Participants will be coded as "yes" (coded as 1) for correctly identifying beverages high in added sugar if they answer all 6 questions correctly.
Thinking about harms of sugary drinks | Assessed once a week for up to 4 weeks, starting on the day of enrollment.
  Measured using 1 survey item: "How much did the labels make you think about the health problems caused by sugary drinks?" The 5-point response scale ranges from "Not at all" (coded as 1) to "A great deal" (coded as 5). Higher scores indicate greater thinking about harms of sugary drinks.
Perceived healthfulness of sugary drinks | Assessed once a week for up to 4 weeks, starting on the day of enrollment.
  Measured using 1 survey item: "How healthy or unhealthy are sugary drinks?" The 5-point response scale ranges from "Very unhealthy" (coded as 1) to "Very healthy" (coded as 5). Higher scores indicate greater perceived healthfulness of sugary drinks.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Hall, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Lindsey Smith Taillie, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT07294053/Prot_SAP_001.pdf